CLINICAL TRIAL: NCT05668975
Title: The Effects of Inspiratory Muscle Training on Diaphragm Thickness, Inspiratory Muscle Strength and Exercise Capacity in Individuals With Sarcopenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Eren Özdoğan, Physiotherapist, MSc Student in Exercise Physiology, Istanbul University, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ErenOzdogan-001
Record Dates: First submitted 2022-11-17; First posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Sarcopenia
Keywords: Inspiratory Muscle Training; Diaphragm Thickness; Respiratory Sarcopenia; Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group (Experimental): Individuals with sarcopenia in this group will perform three sets of 10 repetitions, with 1-minute of rest allocated between sets, twice daily, 5 days per week for eight weeks. The first session will be performed supervised in a clinic, other sessions will be performed at home. Telephone contact will be held twice a week to ensure the completion of training and clarify any doubts. Training intensity will be set at 60% of the maximum inspiratory pressure for the first week then will be set at %70 of the maximum inspiratory pressure for the second week. After the second week, training intensity will be increased as much as participants tolerated at the start of each week.
  Interventions: Device: Inspiratory Muscle Training
- Sham Group (Sham Comparator): Individuals with sarcopenia in this group will perform two sets of 10 repetitions, with 1-minute of rest allocated between sets, one time a day, 2 days per week for eight weeks. The first session will be performed supervised in a clinic, other sessions will be performed at home. Training intensity will be set at 10 cm H₂O for all training sessions.
  Interventions: Device: Inspiratory Muscle Training

INTERVENTIONS:
Device: Inspiratory Muscle Training — A mechanical pressure threshold loading device (POWERbreathe, POWERbreathe International Ltd, UK) will be used for the training.

SUMMARY:
Sarcopenia, according to EWGSOP2(European Working Group on Sarcopenia in Older People-2019), is a progressive and generalised skeletal muscle disorder that is associated with increased likelihood of adverse outcomes including falls, fractures, physical disability, and mortality. Changes in muscle strength and muscle mass that occur with aging are not only limited to the skeletal muscles surrounding the axial and appendicular skeleton, but also occur in the respiratory muscles. With aging, respiratory muscle strength decreases, muscle mass decreases, and respiratory functions decline. In sarcopenic individuals; maximum inspiratory pressure (MIP), maximum expiratory pressure (MEP) and diaphragm muscle thickness values were found to be significantly lower.

It is known that exercise is the most effective and valid way to treat sarcopenia. Considering the positive effects of IMT (Inspiratory Muscle Training) on both respiratory and physical parameters in the elderly population, we think that these changes can also be observed in sarcopenic individuals. Therefore, the aim of this study is to investigate the effects of inspiratory muscle training on diaphragm thickness, inspiratory muscle strength, and exercise capacity in sarcopenic individuals.

ELIGIBILITY:
Inclusion Criteria:

* People who are diagnosed with confirmed sarcopenia or severe sarcopenia according to EWGSOP2 (European Working Group on Sarcopenia in Older People-2019)
* Getting a score of 24 or higher on the mini-mental state test

Exclusion Criteria:

* Presence of chronic lung and/or cardiovascular disease
* Presence of severe orthopedic diseases which may affect participants' mobility
* Presence of uncontrollable hypertension and/or diabetes.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-12 (Actual); Primary Completion 2023-01-15 (Estimated); Study Completion 2023-02-05 (Estimated)

PRIMARY OUTCOMES:
Maximal Inspiratory Pressure | Eight weeks
  Maximal inspiratory pressure (MIP) will be measured using an electronic mouth pressure device (Micro RPM). At least 3 repetitions will be performed and the measurement will be repeated until there is less than a 5% difference between the best and the second-best measurement.
Diaphragm Thickness Measurement at Quiet Breathing | Eight weeks
  Diaphragm thickness measurement will be performed with the Toshiba Aplio 500 ultrasound device at Istanbul University, Istanbul Faculty of Medicine, Department of Sports Medicine. Diaphragm thickness will be measured as the vertical distance between the pleural and peritoneal layer at quiet breathing. Measurement will be performed on the right hemidiaphragm with the volunteer in the supine position. The measurement will be performed 3 times and the average value will be calculated. The value will be expressed in millimeters (mm).
Diaphragm Thickness Measurement at Total Lung Capacity (TLC) | Eight weeks
  Diaphragm thickness measurement will be performed with the Toshiba Aplio 500 ultrasound device at Istanbul University, Istanbul Faculty of Medicine, Department of Sports Medicine. Diaphragm thickness will be measured as the vertical distance between the pleural and peritoneal layer at Total Lung Capacity (TLC). Measurement will be performed on the right hemidiaphragm with the volunteer in the supine position. The measurement will be performed 3 times and the average value will be calculated. The value will be expressed in millimeters (mm).
Diaphragm Thickness Measurement at Functional Residual Capacity (FRC) | Eight weeks
  Diaphragm thickness measurement will be performed with the Toshiba Aplio 500 ultrasound device at Istanbul University, Istanbul Faculty of Medicine, Department of Sports Medicine. Diaphragm thickness will be measured as the vertical distance between the pleural and peritoneal layer at Functional Residual Capacity [FRC]. Measurement will be performed on the right hemidiaphragm with the volunteer in the supine position. The measurement will be performed 3 times and the average value will be calculated. The value will be expressed in millimeters (mm).
Diaphragm Elastography Measurement at Quiet Breathing | Eight weeks
  Diaphragm elastography measurement will be performed with the Toshiba Aplio 500 ultrasound device at Istanbul University, Istanbul Faculty of Medicine, Department of Sports Medicine. The measurement will be performed on the right hemidiaphragm with the volunteer in the supine position. The measurement will be performed 2 times and the average value will be calculated. The value will be expressed in kPa (kilopascal).
Diaphragm Elastography Measurement at Total Lung Capacity (TLC) | Eight weeks
  Diaphragm elastography measurement will be performed with the Toshiba Aplio 500 ultrasound device at Istanbul University, Istanbul Faculty of Medicine, Department of Sports Medicine. The measurement will be performed on the right hemidiaphragm with the volunteer in the supine position. The measurement will be performed 2 times and the average value will be calculated. The value will be expressed in kPa (kilopascal).
Diaphragm Elastography Measurement at Functional Residual Capacity (FRC) | Eight weeks
  Diaphragm elastography measurement will be performed with the Toshiba Aplio 500 ultrasound device at Istanbul University, Istanbul Faculty of Medicine, Department of Sports Medicine. The measurement will be performed on the right hemidiaphragm with the volunteer in the supine position. The measurement will be performed 2 times and the average value will be calculated. The value will be expressed in kPa (kilopascal).
Exercise Capacity Measurement | Eight weeks
  The exercise capacity of the participants will be evaluated with six-minute walk test (6MWT).

SECONDARY OUTCOMES:
Pulmonary Function Test [Forced Vital Capacity (FVC)] | Eight weeks
  The pulmonary function test [Forced Vital Capacity (FVC)] will be performed with Spirobank Mir (SN A23-048) / Winspro v.3.1.1 open circuit spirometer.
Pulmonary Function Test [Forced Expiratory Volume in the first second (FEV1)] | Eight weeks
  The pulmonary function test [Forced Expiratory Volume in the first second (FEV1)] will be performed with Spirobank Mir (SN A23-048) / Winspro v.3.1.1 open circuit spirometer.
Pulmonary Function Test [Peak Expiratory Flow Rate (PEFR)] | Eight weeks
  The pulmonary function test [Peak Expiratory Flow Rate (PEFR)] will be performed with Spirobank Mir (SN A23-048) / Winspro v.3.1.1 open circuit spirometer.
Pulmonary Function Test [Forced expiratory flow 25-75 (FEF25-75%)] | Eight weeks
  The pulmonary function test [Forced expiratory flow 25-75 (FEF25-75%)] will be performed with Spirobank Mir (SN A23-048) / Winspro v.3.1.1 open circuit spirometer.
Assesment of Quality of Life | Eight weeks
  Participants' quality of life will be assessed by the Sarcopenia and Quality of Life (SarQoL) questionnaire. The highest score is 100 and a higher score indicates a better level of quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Üniversitesi İstanbul Tıp Fakültesi Spor Hekimliği Anabilim Dalı, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Ohara DG, Pegorari MS, Oliveira Dos Santos NL, de Fatima Ribeiro Silva C, Monteiro RL, Matos AP, Jamami M. Respiratory Muscle Strength as a Discriminator of Sarcopenia in Community-Dwelling Elderly: A Cross-Sectional Study. J Nutr Health Aging. 2018;22(8):952-958. doi: 10.1007/s12603-018-1079-4. PMID 30272099
- [Background] Deniz O, Coteli S, Karatoprak NB, Pence MC, Varan HD, Kizilarslanoglu MC, Oktar SO, Goker B. Diaphragmatic muscle thickness in older people with and without sarcopenia. Aging Clin Exp Res. 2021 Mar;33(3):573-580. doi: 10.1007/s40520-020-01565-5. Epub 2020 May 13. PMID 32406014
- [Background] Souza H, Rocha T, Pessoa M, Rattes C, Brandao D, Fregonezi G, Campos S, Aliverti A, Dornelas A. Effects of inspiratory muscle training in elderly women on respiratory muscle strength, diaphragm thickness and mobility. J Gerontol A Biol Sci Med Sci. 2014 Dec;69(12):1545-53. doi: 10.1093/gerona/glu182. PMID 25395284